CLINICAL TRIAL: NCT05763030
Title: Sleep Promotion Intervention for Preschool Children in Bangladesh
Brief Title: Sleep Promotion Intervention in Bangladesh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Ayesha Sania, Associate Research Scientist, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAU7943; 1K01TW012425-01 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Sleep
Keywords: Sleep health; Sleep promotion; Child sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parent questionnaires and sleep characteristics of children (actigraphy and parent report) will be collected at three-time points- Time 1, 2, and 3. Time 1 is the first Baseline Data Collection for the Control Group and Intervention Group, and these data will be collected before the intervention group starts the 3-week intervention. Between Time 1 and Time 2, the Intervention Group will receive the 3-week intervention at the childcare center.
  Interventions: Behavioral: Adapted Sleep Well, Bee Well (SWBW)
- Control (No Intervention): The control arm will not receive the intervention. They will be assessed at time 1 and again at 2, following the completion of intervention in the intervention arm

INTERVENTIONS:
Behavioral: Adapted Sleep Well, Bee Well (SWBW) — The SWBW is a 3-week multilevel behavioral sleep intervention that targets organizational (daycare worker-parent), interpersonal (parent-child, daycare worker-child), and individual (child) levels. It provides parent education supporting parent-child interaction at bedtime, helps to adopt a bedtime routine and early bedtime (Table 4). At the beginning of the 3-week intervention period, the parent and teacher co-develop tailored sleep health goals towards meeting the Bedtime, Environment, and Duration (BED) recommendations139-141 for the child. Parents receive an inexpensive bedtime kit, a storybook, and an informational brochure. The parent and child select four activities from the kit to perform at bedtime every night. The brochure has a section for the parents to write sleep goals. During the intervention, daycare teachers provide daily feedback support to parents at pick-up or drop-off. The program has a manualized structured curriculum suitable for use by paraprofessionals.
  Arms: Intervention

SUMMARY:
Using a pragmatic cluster randomized trial, this study aims to examine the feasibility and acceptability of a 3-week behavioral sleep intervention and to test the preliminary efficacy of the intervention compared to a wait-list control with children ages 2-3 years old at two Early Learning Centers on preschooler's sleep health in Dhaka, Bangladesh.

The investigators will use novel, inexpensive wearable technology to measure sleep health of children at ages 2, 3, and 4 years in a total of 60 families of 2-3 year-old healthy children and teachers from both childcare centers. The program teaches early childhood educators about healthy sleep for young children and will train them to be confident facilitators of educational conversations about sleep with parents.

Parent questionnaires and sleep characteristics of children (actigraphy and parent report) will be collected at three-time points- Time 1, 2, and 3. Time 1 is the first Baseline Data Collection for the Control Group and Intervention Group, and these data will be collected before either group starts the 3-week intervention. Between Time 1 and Time 2, the Intervention Group will receive the 3-week intervention at the childcare center. Time 2 data collection for both groups will occur during the week following the completion of the intervention received by the Intervention Group. Time 2 data will serve as post-intervention data for the Intervention Group.

DETAILED DESCRIPTION:
Poor sleep in children is a growing public health concern worldwide. Sleep health is a multidimensional construct (sleep-related behaviors, satisfaction, alertness, timing, efficiency, and duration) influenced by a complex interplay of social-ecological factors. Sleep impacts a range of physical health and neurodevelopmental outcomes including children's executive function (EF), growth, and obesity risk, which are public health priorities in low-and-middle-income countries (LMICs). Early EFs are predictive of social competence and academic performance and economic achievement in later life. Childhood obesity is a rapidly growing health issue in LMICs and a leading risk factor of diabetes. Interventions targeting modifiable sleep behavior have the potential to improve long-term physical and neurodevelopmental outcomes for millions of children in LMICs. Most data on children's sleep health are from high-income settings, and the recommendations based on these studies are not directly relevant to LMICs. Emerging evidence shows multiple cross-cultural differences in sleep dimensions in early childhood. Children in Asian countries have a significantly later bedtime and shorter sleep duration compared to children in Western countries. Recent research and our preliminary data suggest that 40% of preschool children in urban Bangladesh sleep less than the recommended duration (10-13 hours) by the World Health Organization (WHO). Evidence from high-income settings links individual (e.g., age, screen time, physical activity), interpersonal (e.g., maternal mood, parenting stress, mother-child interaction), and social (e.g., social socioeconomic condition, household crowding) factors to childhood sleep. We aim to study the determinants of sleep health using a socioecological framework, and the role of sleep health on growth and neurodevelopmental outcomes among 300 preschool children in Bangladesh, a lower-middle-income country in South Asia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 2-3 years
* Attending early learning centers

Exclusion Criteria:

* Diagnosed with cerebral palsy, severe developmental delay, cardiac disease, or autism
* Known to be born preterm or low birth weight.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2027-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility and acceptability | 21 days
  To determine the feasibility and acceptability of the intervention among families of 2-3 years healthy children and teachers, data will be collected using study-specific Likert-scale surveys. Biweekly site visits and recorded field notes on fidelity will be collected. Together, these field notes will assist in determining the need for intervention refinement and standardization of the intervention manual in preparation for a larger, full-scale future trial.
  The feasibility goals include >50% enrollment and >80% retention rates. Approximate time to complete: 10 minutes. This will be collected at the end of the intervention. The investigators anticipate that the program will be acceptable and feasible to the early learning centers, teachers, and parents.
Change in Parental knowledge and beliefs about children's sleep | 21 days
  Knowledge, attitudes, self-efficacy, and beliefs about sleep in children (KASB) will be administered. There are seven self-efficacy items. The survey will be collected at Time 1, 2, and 3. The score ranges from 0-76. The investigators anticipate that parental knowledge, attitudes, self-efficacy, and beliefs about their children's sleep will improve upon completion of the intervention.

SECONDARY OUTCOMES:
Change in Children's bedtime. | 21 days
  The bedtime sleep characteristics will be measured with the Respironics Actiwatch (AW2), an accelerometer placed on child's wrist. Reliability for actigraphy in preschool children ranges from .67-.85 when measuring sleep duration. The children will wear the water resistant Actiwatch 2 for seven 24-hour periods at Time 1, 2, and 3. The investigators hypothesize that the intervention will improve children' objectively measured bedtime (goal: bedtime before 9:00PM or at least 45 minutes earlier from baseline). Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Bedtime Variability | 21 days
  Night-to-night variability of bedtime will be calculated using a series of successive differences created by calculating the differences among adjacent observations within the same subject from the Actiwatch 2 data at Time 1, 2, and 3. The mean squared successive differences (MSSD) can be used to compute the MSSD that is considered to be an index of variability/instability. The investigators hypothesize that the intervention will improve children' objectively measured bedtime variability. Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Children's sleep duration. | 21 days
  The sleep characteristic of sleep duration will be measured with the Respironics Actiwatch AW2, an accelerometer placed on the ankle of the children. Reliability for actigraphy in children ranges from .67-.85 when measuring sleep duration. The child will wear the water resistant Actiwatch 2 for seven 24-hour periods at Time 1, 2, and 3. The investigators hypothesize that child's sleep duration will increase by 45 minutes after receiving the intervention. Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Children's Sleep Duration Variability | 21 days
  Night-to-night variability of sleep duration will be calculated using a series of successive differences created by calculating the differences among adjacent observations within the same subject from the Actiwatch 2 data at Time 1, 2, and 3. The mean squared successive differences can be used to compute the MSSD that is considered to be an index of variability/instability. The investigators hypothesize that the intervention will improve children's objectively measured sleep duration variability. Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Bedtime Routine | 21 days
  Parent reported sleep characteristics will be measured with the Brief Infant Sleep Questionnaire-Revised (BISQ-R) at Time 1, 2, and 3. Each BISQ-R subscale and total score are scaled from 0 to 100. The BISQ-R has been validated against sleep diaries and actigraphy to elicit parent reports of children's sleep patterns (daytime and nocturnal sleep duration, frequency of awakening, sleep latency), sleep habits [sleeping arrangements, parent-child interactions about sleep (e.g., bedtime behaviors, behaviors related to nocturnal awakenings)], sleep difficulty (i.e., bedtime resistance, nocturnal awakenings, and snoring, a risk factor for sleep apnea]. Questions include information about bedtime routine activities and consistency. Approximate time to complete: 10 minutes. The investigators anticipate an improvement in the three subscales and total score of the parent-reported sleep characteristics after receiving the intervention.
Change in Parent reported sleep characteristics | 21 days
  Parent reported sleep characteristics will be measured with the Brief Infant Sleep Questionnaire-Revised (BISQ-R) at Time 1, 2, and 3. Each BISQ-R subscale and total score are scaled from 0 to 100. The BISQ-R has been validated against sleep diaries and actigraphy to elicit parent reports of children's sleep patterns (daytime and nocturnal sleep duration, frequency of awakening, sleep latency), sleep habits [sleeping arrangements, parent-child interactions about sleep (e.g., bedtime behaviors, behaviors related to nocturnal awakenings)], sleep difficulty (i.e., bedtime resistance, nocturnal awakenings, and snoring, a risk factor for sleep apnea]. Approximate time to complete: 10 minutes. The investigators anticipate an improvement in the total score of the parent-reported sleep characteristics after receiving the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Sania, ScD, Principal Investigator — Columbia University
Locations (1):
- International Centre for Diarrhoeal Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No